CLINICAL TRIAL: NCT06248515
Title: A Phase II Parallel Arm Study of SACITUZUMAB GOVITECAN-HZIY in Patients With Advanced Thymoma and Thymic Carcinoma
Brief Title: A Phase II Trial of Sacituzumab Govitecan in Patients With Advanced Thymic Epithelial Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00007501
Record Dates: First submitted 2024-01-31; First posted 2024-02-08 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Thymoma; Thymic Carcinoma
MeSH Terms: conditions — Thymoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sacituzumab (Experimental)
  Interventions: Drug: Sacituzumab govitecan-hziy

INTERVENTIONS:
Drug: Sacituzumab govitecan-hziy — 10 mg/kg once weekly on Days 1 and 8 of continuous 21-day treatment cycles

SUMMARY:
The goal of this clinical trial is to study the effect of sacituzumab govitecan-hziy in adult patients with advanced thymoma and thymic carcinoma after progressing on at least one prior line of therapy.

The main question it aims to answer is:

• What is the overall response rate (ORR) in patients with advanced thymoma and thymic carcinoma?

Participants will:

* receive a fixed dose of 10 mg/kg given intravenously, once weekly on Days 1 and 8 of continuous 21-day treatment cycles until disease progression or unacceptable toxicity
* have regular blood tests, scans, and examinations to monitor their health.
* have blood and a biopsy of their tumor for research purposes.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 18 years at time of signing informed consent form (ICF)
* Ability to understand and the willingness to sign a written informed consent document
* Patients with histologically confirmed advanced thymoma or thymic carcinoma
* Patients who have experienced disease progression after treatment with at least one prior systemic therapy
* Measurable disease per RECIST v1.1
* Availability of pre-treatment tumor tissue (archival or fresh); If archival tissue is not available and a fresh biopsy is not considered safe and medically feasible by the Investigator, the patient may be approved for enrollment after consultation with the Principal Investigator
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2
* Adequate hematologic and end-organ function, defined by the following laboratory test results, obtained within 14 days prior to initiation of study treatment:
* Absolute neutrophil count (ANC) >/= 1.5 x 10^9/L (1500/uL) without filgrastim support
* Platelet count >/= 100 x 10^9/L (100,000/uL) without transfusion
* Hemoglobin (Hgb) >/= 80 g/L (8 g/dL). Patients may be transfused to meet this criterion.
* Aspartate aminotransferase (AST), alanine transaminase (ALT), and alkaline phosphatase (ALP) </= 2.5 x upper limit of normal (ULN), with the following exceptions:

  * Patients with documented liver metastases: AST and ALT </= 5 x ULN
  * Patients with documented liver or bone metastases: ALP </= 5 x ULN Serum bilirubin </= 1.5 x ULN with the following exception: patients with known Gilbert disease: serum bilirubin </= 3 x ULN
* Creatinine clearance >/= 30 mL/min (calculated using the Cockcroft-Gault formula, see Appendix 2)
* For patients not receiving therapeutic anticoagulation: INR and aPTT </= 1.5 x ULN
* Patients with human immunodeficiency virus (HIV) on effective anti-retroviral therapy with undetectable viral load are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable or on suppressive therapy, if indicated. Patients with a history of hepatitis C virus (HCV) infection must have been treated. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
* Patients with prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods, and agreement to refrain from donating eggs, as defined below:

  * Women must remain abstinent or use contraceptive methods with a failure rate of < 1% per year during the treatment period and for 6 months after the final dose of study treatment. Women must refrain from donating eggs during this same period.
  * A woman is considered to be of childbearing potential if she is postmenarchal, has not reached a postmenopausal state (>/= 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus). The definition of childbearing potential may be adapted for alignment with local guidelines or requirements.
  * Examples of contraceptive methods with a failure rate of > 1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices.
  * The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not adequate methods of contraception.
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm, as defined below:

  * With a female partner of childbearing potential who is not pregnant, men who are not surgically sterile must remain abstinent or use a condom plus an additional contraceptive method that together result in a failure rate of < 1% per year during the treatment period and for 90 days after the final dose of sacituzumab govitecan-hziy. Men must refrain from donating sperm during this this same period.
  * With a pregnant female partner, men must remain abstinent or use a condom during the treatment period and 90 days after the final dose of sacituzumab govitecan-hziy to avoid potential exposure to the embryo.
  * The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not adequate methods of contraception.

Exclusion Criteria:

* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that, in the view of the investigator, contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the patient at high risk from treatment complications.
* Pregnancy or breastfeeding, or intention of becoming pregnant during study treatment or within 6 months after the final dose of study treatment.
* Symptomatic brain metastasis requiring corticosteroids. Patients with treated brain metastases are eligible.
* No concurrent therapy with approved or investigational anticancer therapeutics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-04-25 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | 1 year
  Objective response is defined a confirmed overall response of complete response (CR) or partial response (PR) as assessed by RECIST v1.1. The objective response rate (ORR) will be estimated number of evaluable patients with a documented objective response divided by the total number of evaluable patients.

SECONDARY OUTCOMES:
Duration of response (DOR) | 1 year
  DOR will be evaluated in evaluable patients who had a documented objective response. This is the time from the documented objective response, as assessed by RECIST v1.1, until disease progression or death, whichever occurs first. Patients who are alive without a documented disease progression will be censored at the time of their last disease evaluation.
Progression-free survival (PFS) | 1 year
  Progression-free survival (PFS) is defined as the time from the time of treatment initiation until disease progression or death, whichever occurs first. Patients who are alive without a documented progression will be censored at the time of their last disease evaluation
Overall survival (OS) | 1 year
  Overall survival (OS) is defined as the time of treatment initiation until death. Patients who are alive will be censored at the time of their last contact.

CONTACTS AND LOCATIONS:
Overall Officials: Chul Kim, MD, Principal Investigator — Chul.Kim@gunet.georgetown.edu
Locations (4):
- United States (4):
  - Stanford Cancer Institute, Palo Alto, California
  - Lombardi Comprehensive Cancer Center, Georgetown University, Washington D.C., District of Columbia
  - University of Chicago Medical Center, Chicago, Illinois
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey

IPD SHARING:
Plan to Share IPD: No